CLINICAL TRIAL: NCT03896698
Title: Feasibility Study of Transcranial Ultrasound Stimulation on Alzheimer's Disease Patients
Acronym: TUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Feng-Yi Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: TUS01
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Transcranial Ultrasound Stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TUS treatment (Experimental): AD patients with TUS treatment
  Interventions: Device: Transcranial Ultrasound Stimulation
- Non-TUS treatment (No Intervention): AD patients with Non-TUS treatment

INTERVENTIONS:
Device: Transcranial Ultrasound Stimulation — TUS activate the brain cells
  Arms: TUS treatment

SUMMARY:
Currently, the main treatment method for Alzheimer's disease (AD) is chemotherapy. However, the effectiveness of drugs is moderate and there are several side effects. In this clinical trial, the investigators would like to activate the brain by the transcranial ultrasound stimulation (TUS). This is a feasibility study to evaluate the safety and initial effectiveness of TUS for the treatment of patients with mild AD.

DETAILED DESCRIPTION:
The purpose of this study is to verify the feasibility of low intensity transcranial ultrasound stimulation (TUS) for patients with mild Alzheimer's disease (AD). As a secondary aim, the investigators will explore whether the TUS is associated with improvement in cognitive functioning six and forty-six weeks following the intervention.

Subjects will be randomly assigned to one of two experimental groups which with or without the TUS administration.

The investigators will study up to 20 subjects with mild AD. Initially, subjects will undergo a screening assessment with a study physician to determine medical and psychiatric history, establish AD diagnosis, and undergo a bold draw. Subjects that meet criteria and agree to participate in the study will undergo a follow-up visit. In the baseline measurement visit, participants will first undergo neuropsychological testing. Participants will be randomly assigned to one of two groups. Participants will then be administrated TUS treatment for six weeks. Subsequently, participants will undergo a series of neuropsychological test. A final follow-up assessment will be administered at forty-six weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 55 and 90 years old
2. Weight greater than 50 kg
3. Male or Female
4. Good understanding of written and verbal Chinese
5. Geriatric Depression Scale (GDS) score of < 8
6. Mild AD patients (Mini-Mental State Examination (MMSE) 20-26)
7. Probable AD consistent with NIA/AA criteria
8. The blood flow of bilateral middle cerebral artery M1 can be detected by Transcranial Color Doppler (TCD)
9. Caregiver spending at least 10 hours per week with the patient
10. Agreement to obey the rules of this study
11. Use of cholinesterase inhibitors for AD (Aricept, Namenda, etc.) will be allowed as long as the participant has been on a stable dose for at least six months
12. Does have a reliable caregiver in frequent contact with the patient and can accompany the patient to the clinic and treatment

Exclusion Criteria:

1. Evidence of any other major neurologic or other physical illness that could produce cognitive deterioration, except for mild cognitive impairment (MCI) and any history of stroke or diabetes
2. History of myocardial infarction within the previous year or unstable cardiac disease
3. Any contraindications to MRI scanning such as metallic implants, claustrophibia or too large for MRI scanner
4. History of liver disease or severely impaired renal function
5. The blood flow of either unilateral middle cerebral artery M1 can't be detected by Transcranial Color Doppler (TCD)
6. Major psychiatric disorders, such as bipolar disorder or schizophrenia, or persons with current untreated major depression
7. Pregnant or breastfeeding women

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Device and procedure related adverse events recording | up to 46 weeks after treatment
  Rate of adverse events following each treatment through end of study Clinical and MRI evaluation

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | Change from baseline at 7, 12, 24, and 52 week
  ADAS was designed to measure the severity of the most important symptoms of Alzheimer's disease (AD). Its subscale ADAS-cog is the most popular cognitive testing instrument used in clinical trials of nootropics. It consists of 11 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD. The test administrator adds up points for the errors in each task of the ADAS-Cog for a total score. Total scores range from 0-70. The greater the dysfunction, the greater the score.
Clinical Dementia Rating (CDR) | Change from baseline at 12 and 52 week
  The Clinical Dementia Rating or CDR is a numeric scale used to quantify the severity of symptoms of dementia (i.e. its 'stage'). Using a structured-interview protocol, qualified health professional assesses a patient's cognitive and functional performance in six areas: memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care. Scores in each of these are combined to obtain a composite score ranging from 0 through 3, with 0 meaning of no symptoms, 0.5 very mild dementia, 1 mild dementia, 2 moderate dementia and 3 severe dementia.
Neuropsychiatric Inventory Questionnaire (NPI-Q) | Change from baseline at 12 and 52 week
  NPI-Q is a carer-based tool that assesses the possible presence of 12 symptoms in dementia cases, including delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, night-time behavioral disturbances and appetite/eating disturbances. The severity scale has scores ranging from 1 to 3 points (1=mild; 2=moderate; and 3=severe) and the scale for assessing caregiver distress has scores ranging from 0 to 5 points (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=extreme distress). The total scores of severity and caregiver stress are summed of each 12 items separately, with with higher scores indicating a greater number of neuropsychiatric symptoms or distress.
Transcranial Doppler (TCD) | Changes in blood flow from baseline at 12 and 52 week
  Cerebral blood flow evaluation
Magnetic Resonance Image (MRI) | Change from baseline at 12 and 52 week
  Brain observation

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Yi Yang, Ph.D., Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Chen TT, Lan TH, Yang FY. Low-Intensity Pulsed Ultrasound Attenuates LPS-Induced Neuroinflammation and Memory Impairment by Modulation of TLR4/NF-kappaB Signaling and CREB/BDNF Expression. Cereb Cortex. 2019 Apr 1;29(4):1430-1438. doi: 10.1093/cercor/bhy039. PMID 30873554
- [Background] Chen CM, Wu CT, Yang TH, Liu SH, Yang FY. Preventive Effect of Low Intensity Pulsed Ultrasound against Experimental Cerebral Ischemia/Reperfusion Injury via Apoptosis Reduction and Brain-derived Neurotrophic Factor Induction. Sci Rep. 2018 Apr 3;8(1):5568. doi: 10.1038/s41598-018-23929-8. PMID 29615782
- [Background] Chen SF, Su WS, Wu CH, Lan TH, Yang FY. Transcranial Ultrasound Stimulation Improves Long-Term Functional Outcomes and Protects Against Brain Damage in Traumatic Brain Injury. Mol Neurobiol. 2018 Aug;55(8):7079-7089. doi: 10.1007/s12035-018-0897-z. Epub 2018 Jan 30. PMID 29383687
- [Background] Su WS, Wu CH, Chen SF, Yang FY. Low-intensity pulsed ultrasound improves behavioral and histological outcomes after experimental traumatic brain injury. Sci Rep. 2017 Nov 14;7(1):15524. doi: 10.1038/s41598-017-15916-2. PMID 29138458
- [Background] Su WS, Wu CH, Chen SF, Yang FY. Transcranial ultrasound stimulation promotes brain-derived neurotrophic factor and reduces apoptosis in a mouse model of traumatic brain injury. Brain Stimul. 2017 Nov-Dec;10(6):1032-1041. doi: 10.1016/j.brs.2017.09.003. Epub 2017 Sep 7. PMID 28939348
- [Background] Huang SL, Chang CW, Lee YH, Yang FY. Protective Effect of Low-Intensity Pulsed Ultrasound on Memory Impairment and Brain Damage in a Rat Model of Vascular Dementia. Radiology. 2017 Jan;282(1):113-122. doi: 10.1148/radiol.2016160095. Epub 2016 Jul 11. PMID 27399328
- [Background] Liu SH, Lai YL, Chen BL, Yang FY. Ultrasound Enhances the Expression of Brain-Derived Neurotrophic Factor in Astrocyte Through Activation of TrkB-Akt and Calcium-CaMK Signaling Pathways. Cereb Cortex. 2017 Jun 1;27(6):3152-3160. doi: 10.1093/cercor/bhw169. PMID 27252349
- [Background] Su WS, Tsai ML, Huang SL, Liu SH, Yang FY. Controllable permeability of blood-brain barrier and reduced brain injury through low-intensity pulsed ultrasound stimulation. Oncotarget. 2015 Dec 8;6(39):42290-9. doi: 10.18632/oncotarget.5978. PMID 26517350
- [Background] Lin WT, Chen RC, Lu WW, Liu SH, Yang FY. Protective effects of low-intensity pulsed ultrasound on aluminum-induced cerebral damage in Alzheimer's disease rat model. Sci Rep. 2015 Apr 15;5:9671. doi: 10.1038/srep09671. PMID 25873429
- [Background] Yang FY, Lu WW, Lin WT, Chang CW, Huang SL. Enhancement of Neurotrophic Factors in Astrocyte for Neuroprotective Effects in Brain Disorders Using Low-intensity Pulsed Ultrasound Stimulation. Brain Stimul. 2015 May-Jun;8(3):465-73. doi: 10.1016/j.brs.2014.11.017. Epub 2014 Dec 4. PMID 25558041